CLINICAL TRIAL: NCT00877877
Title: Follow-up Study to Evaluate the Long-term Immunogenicity and Safety of a HPV Vaccine (GSK 580299) in Healthy Female Subjects
Brief Title: Evaluation of Long-term Immunogenicity and Safety of a Human Papillomavirus (HPV) Vaccine in Healthy Female Subjects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 111375; 2008-000369-44 (EudraCT Number)
Record Dates: First submitted 2009-03-26; First posted 2009-04-08 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: Infections, Papillomavirus; Papillomavirus Vaccines
Keywords: HPV vaccine; cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Blood Specimen Collection

ARMS (1):
- Cervarix Group (Other): Subjects in the Cervarix Group of the primary study (NCT00196924), who had then received 3 doses of Cervarix™ vaccine intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6 month vaccination schedule.
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood samples were to be collected at Months 60, 72, 84, 96, 108 and 120

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the necessary cause of cervical cancer. This study is designed to evaluate the long-term immunogenicity and safety of the 580299 HPV vaccine up to 10 years after administration of the first dose of HPV vaccine (Month 0) administered in the primary study 580299/013. This protocol posting deals with objectives & outcome measures of the extension phase from Month 60 to Month 120. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT00196924). The objectives & outcome measures of the extension phase up to Month 48 are presented in a separate protocol posting (NCT00316706).

DETAILED DESCRIPTION:
Subjects were aged 10-14 years at the time of entry into the primary study. No vaccine will be administered in this extension study.

Results on outcome measures describing analyses on other studies are not reported in this record. Please refer to the records mentioned in the respective outcome measure titles.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parents or legally acceptable representative (LAR) can and will comply with the requirements of the protocol should be enrolled in the study.
* A female enrolled in the immunogenicity subset of study 580299-013, who received three doses of HPV vaccine and participated in the extension study of 580299-013.
* Written informed assent obtained from the subject. For subjects below the legal age of consent, written informed consent must be obtained from a parent or legally acceptable representative of the subject.

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Use of any investigational or non-registered product (drug or vaccine) or planned use during the study period.
* Administration or planned administration of any HPV vaccine, other than the vaccine administered in study 580299-013.
* Chronic administration of immunosuppressants or other immune-modifying drugs occurring within the three months preceding study entry.
* Administration of immunoglobulins and/or any blood products occurring within the three months preceding study entry.

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 632 (Actual)
Dates: Start 2009-05-07 (Actual); Primary Completion 2015-01-06 (Actual); Study Completion 2015-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- GSK Investigational Site, Bogotá, Colombia
- Germany (19):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Bützow, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Harrislee, Schleswig-Holstein
  - GSK Investigational Site, Niebüll, Schleswig-Holstein
  - GSK Investigational Site, Weimar, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Tegucigalpa, Francisco Morazán Department, Honduras
- Panama (2):
  - GSK Investigational Site, Arraijan/Vista Alegre, Provincia de Panamá
  - GSK Investigational Site, La Chorrera
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=3315

REFERENCES:
- [Background] Schwarz TF, Huang LM, Lin TY, Wittermann C, Panzer F, Valencia A, Suryakiran PV, Lin L, Descamps D. Long-term immunogenicity and safety of the HPV-16/18 AS04-adjuvanted vaccine in 10- to 14-year-old girls: open 6-year follow-up of an initial observer-blinded, randomized trial. Pediatr Infect Dis J. 2014 Dec;33(12):1255-61. doi: 10.1097/INF.0000000000000460. PMID 24978856
- [Background] Schwarz TF, Huang LM, Valencia A, Panzer F, Chiu CH, Decreux A, Poncelet S, Karkada N, Folschweiller N, Lin L, Dubin G, Struyf F. A ten-year study of immunogenicity and safety of the AS04-HPV-16/18 vaccine in adolescent girls aged 10-14 years. Hum Vaccin Immunother. 2019;15(7-8):1970-1979. doi: 10.1080/21645515.2019.1625644. Epub 2019 Jul 17. PMID 31268383
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 111375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who participated in the primary study (NCT00196924) and received 3 doses of Cervarix.
Pre-assignment Details: Subjects enrolled in this study were primed with Cervarix vaccine as part of study NCT00196924. Subjects not returning for a specific visit were not withdrawn and could participate in the subsequent follow-up phases. Actual enrollment differed depending on the rate of return for the follow-up study, so not all subjects enrolled came to each visit.
Period: Year 5
Arm/Group | Cervarix Group
Started | 397
Completed | 397
Not Completed | 0
Period: Year 6
Arm/Group | Cervarix Group
Started | 529
Completed | 529
Not Completed | 0
Period: Year 7
Arm/Group | Cervarix Group
Started | 523
Completed | 523
Not Completed | 0
Period: Year 8
Arm/Group | Cervarix Group
Started | 522
Completed | 522
Not Completed | 0
Period: Year 9
Arm/Group | Cervarix Group
Started | 507
Completed | 507
Not Completed | 0
Period: Year 10
Arm/Group | Cervarix Group
Started | 495
Completed | 495
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cervarix Group
Number analyzed (Participants) | 529
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Year 5 | 17.1 (1.40)
  Year 6 | 18.0 (1.40)
  Year 7 | 19.0 (1.39)
  Year 8 | 20.0 (1.40)
  Year 9 | 21.1 (1.42)
  Year 10 | 22.0 (1.40)
Sex/Gender, Customized [Number; unit: Participants] — Year 5 cohort
  Participants
    Female | 397
    Male | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Year 6 cohort
  Participants
    Female | 529
    Male | 0
Sex/Gender, Customized [Number; unit: Participants] — Year 7 cohort
  Participants
    Female | 523
    Male | 0
Sex/Gender, Customized [Number; unit: Participants] — Year 8 cohort
  Participants
    Female | 522
    Male | 0
Sex/Gender, Customized [Number; unit: Participants] — Year 9 cohort
  Participants
    Female | 507
    Male | 0
Sex/Gender, Customized [Number; unit: Participants] — Year 10 cohort
  Participants
    Female | 495
    Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects With Anti-HPV-16/18 Antibody Titers Equal to or Above Cut-off Values.
Description: Anti-HPV-16 assay cut-off value was defined as 8 ELISA units per milliliter (EL.U/mL). Anti-HPV-18 assay cut-off value was defined as 7 EL.U/mL.
  Seroconversion was defined as the appearance of antibodies (i.e. titer greater than or equal to the cut-off value) in the serum of subjects seronegative before vaccination.
  A seronegative subject is a subject with antibody titer < 8 or 7 EL.U/mL prior to vaccination.
  A seropositive subject is a subject with antibody titer >= 8 or 7 EL.U/mL prior to vaccination.
Time Frame: At Month 60
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity Month 60 which included all evaluable subjects from the primary study (NCT00196924) for whom serology results were available at the Month 60 blood sampling timepoint.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 358
Subjects
  anti-HPV-16 Month 60 [N=353] | 353
  anti-HPV-18 Month 60 [N=358] | 358

2. Primary Outcome: Number of Seroconverted Subjects With Anti-HPV-16/18 Antibody Titers Equal to or Above Cut-off Values.
Description: as for outcome 1
Time Frame: At Month 72
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity Month 72 which included all evaluable subjects from the primary study (NCT00196924) for whom serology results were available at the Month 72 blood sampling timepoint.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 478
Subjects
  anti-HPV-16 Month 72 [N=475] | 475
  anti-HPV-18 Month 72 [N=478] | 478

3. Primary Outcome: Number of Seroconverted Subjects With Anti-HPV-16/18 Antibody Titers Equal to or Above Cut-off Values.
Description: as for outcome 1
Time Frame: At Month 84
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity Month 84 which included all evaluable subjects from the primary study (NCT00196924) for whom serology results were available at the Month 84 blood sampling timepoint.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 473
Subjects
  HPV-16 Month 84 [N=469] | 469
  HPV-18 Month 84 [N=473] | 473

4. Primary Outcome: Number of Seroconverted Subjects With Anti-HPV-16/18 Antibody Titers Equal to or Above Cut-off Values.
Description: as for outcome 1
Time Frame: At Month 96
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity Month 96 which included all evaluable subjects from the primary study (NCT00196924) for whom serology results were available at the Month 96 blood sampling timepoint.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 477
Subjects
  anti-HPV-16 Month 96 [N=473] | 473
  anti-HPV-18 Month 96 [N=477] | 477

5. Primary Outcome: Anti-human Papillomavirus-16 and 18 (Anti-HPV-16/18) Antibody Titers
Description: Anti-HPV-16 and 18 antibody titers are given in Geometric Mean Titers (GMTs) in Enzyme-linked Immunosorbent Assay (ELISA) Units per milliliter (EL.U/mL).
Time Frame: At Month 60
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group
Number analyzed (Participants) | 376
EL.U/mL
  anti-HPV-16 Month 60 [N=376] | 2262.9 [2069.1 to 2475.0]
  anti-HPV-18 Month 60 [N=376] | 778.6 [703.1 to 862.1]

6. Primary Outcome: Anti-human Papillomavirus-16 and 18 (Anti-HPV-16/18) Antibody Titers
Description: as for outcome 5
Time Frame: At month 72
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group
Number analyzed (Participants) | 502
EL.U/mL
  anti-HPV-16 Month 72 [N=502] | 1973.9 [1827.9 to 2131.6]
  anti-HPV-18 Month 72 [N=502] | 762.8 [701.0 to 830.1]

7. Primary Outcome: Anti-human Papillomavirus-16 and 18 (Anti-HPV-16/18) Antibody Titers
Description: as for outcome 5
Time Frame: At Month 84
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group
Number analyzed (Participants) | 494
EL.U/mL
  anti-HPV-016 Month 84 [N=494] | 1756.7 [1622.7 to 1901.7]
  anti-HPV-018 Month 84 [N=494] | 609.7 [559.0 to 664.9]

8. Primary Outcome: Anti-human Papillomavirus-16 and 18 (Anti-HPV-16/18) Antibody Titers
Description: as for outcome 5
Time Frame: At Month 96
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group
Number analyzed (Participants) | 499
EL.U/mL
  anti-HPV-16 Month 96 [N=499] | 1671.0 [1548.1 to 1803.7]
  anti-HPV-18 Month 96 [N=499] | 679.0 [623.5 to 739.4]

9. Primary Outcome: Number of Seroconverted Subjects With Anti-HPV-16/18 Antibody Titers Equal to or Above Cut-off Values.
Description: as for outcome 1
Time Frame: At Month 108
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity Month 108 which included all evaluable subjects from the primary study (NCT00196924) for whom serology results were available at the Month 108 blood sampling timepoint.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 374
Subjects
  Anti-HPV-16 Month 108 [N=374] | 372
  Anti-HPV-18 Month 108 [N=370] | 368

10. Primary Outcome: Anti-human Papillomavirus-16 and 18 (Anti-HPV-16/18) Antibody Titers
Description: as for outcome 5
Time Frame: At Month 108
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity Month 108 which included all evaluable subjects from the primary study (NCT00196924) for whom serology results were available at the Month 108 blood sampling timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/ML
Arm/Group | Cervarix Group
Number analyzed (Participants) | 392
EL.U/ML
  Anti-HPV-16 Month 108 [N=392] | 1946.5 [1779.7 to 2128.9]
  Anti-HPV-18 Month 108 [N=391] | 754.0 [685.4 to 829.4]

11. Primary Outcome: Anti-human Papillomavirus-16 and 18 (Anti-HPV-16/18) Antibody Titers
Description: as for outcome 1
Time Frame: At Month 120
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity Month 120 which included all evaluable subjects from the primary study (NCT00196924) for whom serology results were available at the Month 120 blood sampling timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group
Number analyzed (Participants) | 416
EL.U/mL
  Anti-HPV-16 Month 120 [N=416] | 1607.9 [1480.8 to 1746.1]
  Anti-HPV-18 Month 120 [N=415] | 608 [552.5 to 669.1]

12. Primary Outcome: Number of Seroconverted Subjects With Anti-HPV-16/18 Antibody Titers Equal to or Above Cut-off Values.
Description: as for outcome 1
Time Frame: At Month 120
Population: as for outcome 11
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 395
Subjects
  Anti-HPV-16 Month 120 [N=393] | 393
  Anti-HPV-18 Month 120 [N=395] | 395

13. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Month 48 to Month 60
Population: The analysis was performed on the Month 60 Total Vaccinated cohort, which included all vaccinated subjects (who had received 3 doses during the primary study (NCT00196924)) for whom data were available for the Month 60 time point.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 397
Subjects | 9

14. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 13
Time Frame: From Month 60 to Month 72
Population: Analysis was performed on the Month 72 Total Vaccinated cohort, which included all vaccinated subjects (who had received 3 doses during the primary study (NCT00196924)) for whom data were available for the Month 72 time point.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 529
Subjects | 20

15. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 13
Time Frame: From Month 72 to Month 84
Population: Analysis was performed on the Month 84 Total Vaccinated cohort, which included all vaccinated subjects (who had received 3 doses during the primary study (NCT00196924)) for whom data were available for the Month 84 time point.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 523
Subjects | 20

16. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 13
Time Frame: From Month 84 to Month 96
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 522
Subjects | 8

17. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 13
Time Frame: From Month 96 to Month 108
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 507
Subjects | 15

18. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 13
Time Frame: From Month 108 to Month 120
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 495
Subjects | 6

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were assessed by time intervals: Months 48-60, Months 60-72, Months 72-84, Months 84-96, Months 96-108 and Months 108-120.
Description: Other (non-serious) Adverse Events were not collected/assessed during this long-term follow-up study.
Groups:
- Cervarix Group From Month 48 Until Month 60: Subjects in the Cervarix Group of the primary study (NCT00196924), who had then received 3 doses of Cervarix™ vaccine intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6 month vaccination schedule and for whom serious adverse events were collected from Month 48 until Month 60.
- Cervarix Group From Month 60 Until Month 72: Subjects in the Cervarix Group of the primary study (NCT00196924), who had then received 3 doses of Cervarix™ vaccine intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6 month vaccination schedule and for whom serious adverse events were collected from Month 60 until Month 72.
- Cervarix Group From Month 72 to Month 84: Subjects in the Cervarix Group of the primary study (NCT00196924), who had then received 3 doses of Cervarix™ vaccine intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6 month vaccination schedule and for whom serious adverse events were collected from Month 72 until Month 84.
- Cervarix Group From Month 84 to Month 96: Subjects in the Cervarix Group of the primary study (NCT00196924), who had then received 3 doses of Cervarix™ vaccine intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6 month vaccination schedule and for whom serious adverse events were collected from Month 84 until Month 96.
- Cervarix Group From Month 96 to Month 108: Subjects in the Cervarix Group of the primary study (NCT00196924), who had then received 3 doses of Cervarix™ vaccine intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6 month vaccination schedule and for whom serious adverse events were collected from Month 96 until Month 108.
- Cervarix Group From Month 108 to Month 120: Subjects in the Cervarix Group of the primary study (NCT00196924), who had then received 3 doses of Cervarix™ vaccine intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6 month vaccination schedule and for whom serious adverse events were collected from Month 108 until Month 120.
Arm/Group | Cervarix Group From Month 48 Until Month 60 | Cervarix Group From Month 60 Until Month 72 | Cervarix Group From Month 72 to Month 84 | Cervarix Group From Month 84 to Month 96 | Cervarix Group From Month 96 to Month 108 | Cervarix Group From Month 108 to Month 120
Serious Adverse Events (participants affected / at risk) | 9/397 | 20/529 | 20/523 | 8/522 | 15/507 | 6/495
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group From Month 48 Until Month 60 (N=397) | Cervarix Group From Month 60 Until Month 72 (N=529) | Cervarix Group From Month 72 to Month 84 (N=523) | Cervarix Group From Month 84 to Month 96 (N=522) | Cervarix Group From Month 96 to Month 108 (N=507) | Cervarix Group From Month 108 to Month 120 (N=495)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 3 | 2 | 1 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skull malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Endometritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Olygohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0
Cerebral cyst (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Congenital megaureter (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Endometritis decidual (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Talipes (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 1
Endometritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.